CLINICAL TRIAL: NCT06106269
Title: Hemorrhoidal Embolization Trial-1 (HEMBO-1)
Brief Title: Outcomes and Quality of Life Following Rectal Artery Embolization for Bleeding Internal Hemorrhoids
Acronym: HEMBO-1
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Terumo Corporation (Industry)
Responsible Party: Principal Investigator, Scott M. Thompson, Principal Investigator, Mayo Clinic
Other Study IDs: 23-002845
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Internal Hemorrhoid
Keywords: Bleeding; Anemia; Hemorrhoid
MeSH Terms: conditions — Hemorrhage; Anemia; Hemorrhoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Rectal Artery Embolization — Subjects will undergo planned rectal artery embolization (RAE) in Vascular and Interventional Radiology per standard clinical protocol.

SUMMARY:
This study will assess how effective and safe rectal artery embolization works to treat symptomatic bleeding predominant internal hemorrhoids.

DETAILED DESCRIPTION:
This is a prospective, single-arm, single center phase I/IIa observational study to systematically investigate outcomes and quality of life in patients with grade II or III bleeding predominant internal hemorrhoids referred to Vascular and Interventional Radiology (VIR) by Colorectal Surgery (CRS) for clinically indicated rectal artery embolization. 20 adult patients who meet the inclusion and exclusion criteria will be consented and enrolled in the study.

During the study, the subject will undergo 6 study visits, one before and five after their clinical rectal artery embolization procedure. Patients referred from the Colorectal Surgery Clinic who are scheduled to undergo rectal artery embolization (RAE) as part of standard clinical care will be enrolled. Baseline anoscopy and clinical evaluation will be performed per standard clinical care in the Colorectal Surgery Clinic and baseline patient reported outcomes and quality of life questionnaires administered. A research pelvis CTA will be performed on a clinical CT scanner per standard clinical imaging protocol for assessment of the rectal arteries prior to embolization. Following rectal artery embolization, subjects will undergo a day 1 post-procedure clinical evaluation in Interventional Radiology followed by repeat anoscopy and clinical evaluation per standard clinical care in the Colorectal Surgery Clinic as well as repeat patient reported outcomes and quality of life questionnaires at 1, 3, 6 and 12 months post rectal artery embolization with a clinical research study coordinator in Vascular and Interventional Radiology, either in person or virtually (video or phone).

The aims of the study are:

Aim 1. To determine the 12-month efficacy of rectal artery embolization with particles + coils for treatment of symptomatic bleeding predominant hemorrhoidal disease

Aim 2. To determine the 12-month safety of rectal artery embolization with particles + coils for treatment of symptomatic bleeding predominant hemorrhoidal disease.

Aim 3. To determine the feasibility of pre-embolization CTA in identifying the hemorrhoidal arteries supplying the hemorrhoidal cushion

ELIGIBILITY:
Inclusion Criteria:

* Grade II or III hemorrhoidal disease as determined by a board-certified colorectal surgeon.
* Persistent or recurrent symptoms following hygiene and dietary measures or medication.
* Bleeding predominant ± pain symptoms.
* Undergoing planned rectal artery embolization (RAE) per standard clinical care.
* Male or female with age greater than 18 years, with the capacity and willingness to provide a written informed consent.
* Negative pregnancy test (if applicable).

Exclusion Criteria:

* Prior hemorrhoid surgery.
* Grade IV hemorrhoidal disease.
* Acute hemorrhoid complications.
* Chronic anal or perianal fissures.
* History of colorectal surgery or pelvic radiation.
* Inflammatory bowel disease.
* Portal hypertension or mesenteric venous congestion/occlusion.
* Inferior mesenteric artery (IMA) or internal iliac artery (IIA) stenosis or occlusion.
* Contraindication to iodinated contrast.
* Pregnant and/or breast-feeding subjects. A negative pregnancy test within 48 hours of the procedure per clinical care.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects referred from the Colon and Rectal Surgery who are scheduled to undergo rectal artery embolization (RAE) as part of their standard clinical care at the Mayo Clinic in Rochester, Minnesota.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in French bleeding score (FBS) | Baseline, 1, 3, 6 and 12 months
  The French bleeding score assesses the intensity of hemorrhoidal bleeding with scores ranging from 0 (no bleeding) to 9 (daily bleeding with anemia requiring blood transfusions)
Adverse Events | Day 1 and 1, 3, 6 and 12 months
  Number of subjects to experience adverse events defined by 1) Common Terminology Criteria for Adverse Events (CTCAE) v6.0, 2) Society of Interventional Radiology [SIR] classifications of postoperative complications and 3) Clavien-Dindo Classification
Diagnostic accuracy of pre-embolization Computed Tomography Angiography (CTA) | Baseline (pre-embolization)
  Diagnostic accuracy and inter-rater agreement of pre-embolization CTA in identifying the hemorrhoidal arteries supplying the hemorrhoidal cushion

SECONDARY OUTCOMES:
Visual Analog Scale (VSS) Pain | Baseline, 1, 3, 6 and 12 months
  Pain values reported by participants will be assessed using a visual analogue scale with a line where each end is marked with "no pain" as 0 on the left, middle with "Moderate pain" as 5, and "worst possible pain" as 10 on the right. Participants will identify their pain level by indicating a point on the line between each end. Pain score 1-3 = mild pain, minimal impact on activities of daily living (ADL's); 4-6 = moderate pain, moderate impact on ADL's; 7-10 = severe pain, major impact on ADL's.
Visual Analog Scale (VAS) for Quality of Life | Baseline, 1, 3, 6 and 12 months
  The quality-of-life score evaluates disease impact with scores ranging from 0 (absence of discomfort) to 4 (permanent discomfort).
Goligher Prolapse Score | Baseline, 1, 3, 6 and 12 months
  The Goligher classification asses the degree of internal hemorrhoid prolapse from I (no prolapse) to IV (irreducible prolapse).
Hemorrhoidal Bleeding Score (HBS) | Baseline, 1, 3, 6 and 12 months
  HBS is sensitive, specific, and reproducible. It can assess the severity of hemorrhoidal bleeding. It also allows quantifying the extent of change in hemorrhoidal bleeding after treatment.
Hemorrhoidal Severity Score (HSS) | Baseline, 1, 3, 6 and 12 months
  The HSS comprises five items. All items included in a domain are scored between 0 and 3 (0 indicating best and 3 worst health status). A total score is obtained by summing the answers to each item. Lower scores indicate better haemorrhoidal health
Vaizey Incontinence Score | Baseline, 1, 3, 6 and 12 months
  The Vaizey incontinence score questionnaire is a seven-item measure in detecting fecal incontinence. The Vaizey consists of seven items, three of which ask about the frequency of incontinence on a 4-point scale ranging from 0 = Never to 4= Daily, followed by a single item about the extent to which symptoms alter lifestyle (using the same 4-point scale). The final three items are concerned with the severity of incontinence using a dichotomous No/Yes response scale (No=0, Yes=2 for items five and six, and 4 for item seven). The Vaizey score is calculated by summing responses across the seven items. A lower score indicates less fecal incontinence (e.g. 0=perfect continence, 24=totally incontinent).
Brief Pain Inventory (BPI) Short Form | Baseline, 1, 3, 6 and 12 months
  The Brief Pain Inventory (BPI) rapidly assesses the severity of pain and its impact on functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Thompson, MD, PhD, Principal Investigator — Mayo Clinic, Vascular and Interventional Radiology; Scott R Kelley, MD, Principal Investigator — Mayo Clinic, Colon and Rectal Surgery
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20556753